CLINICAL TRIAL: NCT01441544
Title: The Effect of Variety on Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 8630B
Record Dates: First submitted 2011-09-25; First posted 2011-09-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Overweight
Keywords: active video games; Energy expenditure
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAREITY (Experimental)
  Interventions: Behavioral: Variety of Active Videogames
- NON-VARIETY (Experimental)
  Interventions: Behavioral: Variety of Active Videogames

INTERVENTIONS:
Behavioral: Variety of Active Videogames — Thirty men and women, aged 18- to 35- years, recruited from the local area, with a normal body mass index (BMI) between 18.5 and 29.9 kg/m, will participate in two experimental sessions, VARIETY (playing the same active video game over 4 sessions) and NON-VARIETY (playing 4 different active video games over 4 sessions), with order of experimental sessions counterbalanced across participants.

SUMMARY:
Increasing physical activity continues to be a challenge among many individuals, particularly those who are overweight. Recent data from the National Health and Nutrition Examination Survey (NHANES) showed that individuals who reported engaging in a variety of activities were more likely to meet national physical activity recommendations compared to those who reported no variety. Incorporating a variety of activities into a physical activity program may be a way to increase physical increase physical activity levels.

One method to increase variety in physical activities is to use active videogames. Videogames that use motion sensors allow a gamer to physically perform a variety of activities. Thus, the purpose ot this laboratory-based investigation is to conduct a study to examine the effect of engaging in a greater variety of active videogames on energy expenditure in 30 non-obese, regularly active adults.

DETAILED DESCRIPTION:
Thirty men and women, aged 18- to 35- years, recruited from the local area, with a normal body mass index (BMI) between 18.5 and 29.9 kg/m, will participate in two experimental sessions, VARIETY and NON-VARIETY, with order of experimental sessions counterbalanced across participants. Participants will be assessed on liking of the active videogames, energy, tiredness, motivation, to succeed, interest in the games, and energy expenditure during the experimental sessions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-25 years are eligible to participate. They will be recruited from flyers posted around campus and in local gyms, and must be willing to participate. They must have a body mass index (BMI) between 18.5 and 29.9 kg/m2.

Exclusion Criteria:

* Participants who have never played an active videogame or are unable to play an active videogame. If the participant dislikes (scoring <50 on a 100 mm visual analogue scale [VAS]) playing the active videogames used in the investigation. Or if the participant engages in less than 150 minutes/week of moderate- to vigorous-intensity physical activity over the previous month.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Energy expenditure in a laboratory session when active videogames are played | End of each session

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, Ph. D, Principal Investigator — University of Tennessee; Dale Bond, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States

REFERENCES:
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] Tudor-Locke C, Brashear MM, Johnson WD, Katzmarzyk PT. Accelerometer profiles of physical activity and inactivity in normal weight, overweight, and obese U.S. men and women. Int J Behav Nutr Phys Act. 2010 Aug 3;7:60. doi: 10.1186/1479-5868-7-60. PMID 20682057
- [Background] Perri MG, Martin AD, Leermakers EA, Sears SF, Notelovitz M. Effects of group- versus home-based exercise in the treatment of obesity. J Consult Clin Psychol. 1997 Apr;65(2):278-85. doi: 10.1037//0022-006x.65.2.278. PMID 9086691
- [Background] Jakicic JM, Winters C, Lang W, Wing RR. Effects of intermittent exercise and use of home exercise equipment on adherence, weight loss, and fitness in overweight women: a randomized trial. JAMA. 1999 Oct 27;282(16):1554-60. doi: 10.1001/jama.282.16.1554. PMID 10546695
- [Background] Otten JJ, Jones KE, Littenberg B, Harvey-Berino J. Effects of television viewing reduction on energy intake and expenditure in overweight and obese adults: a randomized controlled trial. Arch Intern Med. 2009 Dec 14;169(22):2109-15. doi: 10.1001/archinternmed.2009.430. PMID 20008695
- [Background] Jakicic JM, Wing RR, Butler BA, Robertson RJ. Prescribing exercise in multiple short bouts versus one continuous bout: effects on adherence, cardiorespiratory fitness, and weight loss in overweight women. Int J Obes Relat Metab Disord. 1995 Dec;19(12):893-901. PMID 8963358
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Sherwood NE, Jeffery RW. The behavioral determinants of exercise: implications for physical activity interventions. Annu Rev Nutr. 2000;20:21-44. doi: 10.1146/annurev.nutr.20.1.21. PMID 10940325
- [Background] Fitzhugh EC, Thompson DL. Leisure-time walking and compliance with ACSM/AHA aerobic-related physical activity recommendations: 1999-2004 NHANES. J Phys Act Health. 2009 Jul;6(4):393-402. doi: 10.1123/jpah.6.4.393. PMID 19842452
- [Background] Pereira MA, FitzerGerald SJ, Gregg EW, Joswiak ML, Ryan WJ, Suminski RR, Utter AC, Zmuda JM. A collection of Physical Activity Questionnaires for health-related research. Med Sci Sports Exerc. 1997 Jun;29(6 Suppl):S1-205. No abstract available. PMID 9243481
- [Background] Raynor HA, Epstein LH. The relative-reinforcing value of food under differing levels of food deprivation and restriction. Appetite. 2003 Feb;40(1):15-24. doi: 10.1016/s0195-6663(02)00161-7. PMID 12631501
- [Background] Levac D, Pierrynowski MR, Canestraro M, Gurr L, Leonard L, Neeley C. Exploring children's movement characteristics during virtual reality video game play. Hum Mov Sci. 2010 Dec;29(6):1023-38. doi: 10.1016/j.humov.2010.06.006. Epub 2010 Aug 17. PMID 20724014
- [Background] McAuley E, Duncan T, Tammen VV. Psychometric properties of the Intrinsic Motivation Inventory in a competitive sport setting: a confirmatory factor analysis. Res Q Exerc Sport. 1989 Mar;60(1):48-58. doi: 10.1080/02701367.1989.10607413. PMID 2489825
- [Derived] Raynor HA, Cardoso C, Bond DS. Effect of exposure to greater active videogame variety on time spent in moderate- to vigorous-intensity physical activity. Physiol Behav. 2016 Jul 1;161:99-103. doi: 10.1016/j.physbeh.2016.04.016. Epub 2016 Apr 14. PMID 27090231